CLINICAL TRIAL: NCT04425876
Title: A Phase I Study to Assess the Tolerability, Safety and Efficacy of Fluzoparib in Combination With mFOLFIRINOX as Neoadjuvant and Adjuvant Therapy in Patients With Resectable Pancreatic Cancer
Brief Title: A Study of Fluzoparib in Combination With mFOLFIRINOX in Patients With Resectable Pancreatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3162-I-116
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib+mFOLFIRINOX (Experimental): Fluzoparib combined with FOLFIRINOX followed by maintenance Fluzoparib monotherapy
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib combined with mFOLFIRINOX followed by maintenance Fluzoparib monotherapy
  Other Names: SHR3162

SUMMARY:
The study is being conducted to: a) evaluate the tolerability and safety of the co-administration of Fluzoparib and FOLFIRINOX in patients with resectable pancreatic cancer, and establish a maximum tolerated dose and recommended phase II dose of the combination and b) assess the efficacy of the co-administration of Fluzoparib and FOLFIRINOX in patients with resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-79 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
* Expected survival ≥ 6 months.
* Histologically or cytologically confirmed pancreas adenocarcinoma.
* Resectable or borderline resectable pancreatic cancer.
* Adequate organ performance based on laboratory blood tests.
* Presence of at least of one measurable lesion in agreement to RECIST criteria.
* Ability to understand and the willingness to receive a needle biopsy.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had any chemotherapy or radiotherapy prior to entering the study.
* Patients with metastasis disease.
* Previous treatment with a poly ADP-ribose polymerase (PARP) inhibitor.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to oxaliplatin, irinotecan, 5-Fluorouracil or other agents used in the study.
* Previous treatment using CYP3A4 inducers within 3 weeks or inhibitors within 2 weeks.
* Significant cardiovascular disease such as New York Heart Associate Class III/IV, cardiac failure, myocardial infarction, unstable arrhythmia, or evidence of ischemia on ECG within 6 months prior to enrolment.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia.
* Patients with second primary cancer except curatively treated in-situ cancer or slowly progressing malignancy.
* Known active hepatitis B or C infection.
* History of immunodeficiency (including HIV infection) or organ transplantation.
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a dose limited toxicity | 28 Days (first and second cycle)
  Number of participants with a dose limited toxicity
Maximum tolerated dose | Up to 8 months
  Maximum tolerated dose
RP2D | Up to 8 months
  Recommended Phase 2 Dose
R0 resection rate | Up to 2 years
  R0 resection rate of Fluzoparib in combination with FOLFIRINOX as neoadjuvant therapy in patients with resectable pancreatic cancer

SECONDARY OUTCOMES:
AEs | From the first drug administration to within 30 days for the last drug dose
  Incidence of adverse events and associated dose of Fluzoparib
Resection Rate | Up to 2 years
  Resection rate of Fluzoparib in combination with FOLFIRINOX as neoadjuvant therapy in patients with resectable pancreatic cancer
MPR Rate | Up to 2 years
  Major pathological response rate based on central review
Objective response rate | Up to 2 years
  Objective response rate
Disease-free-survival | Up to 2 years
  Disease-free-survival
Event-Free-Survival | Up to 2 years
  Event-Free-Survival
Overall-Survival | Up to 2 years
  Overall-Survival
Minimum concentration (Cmin) | Up to 2 years
  Minimum observed plasma concentration for Fluzoparib

CONTACTS AND LOCATIONS:
Overall Officials: Boyong Shen, M.D., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China